CLINICAL TRIAL: NCT05048771
Title: Fertility and Temporality in Pediatric Oncology
Acronym: FERTITOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Principal Investigator, Isabelle KOSCINSKI, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2019PI269
Record Dates: First submitted 2021-08-25; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Fertility Issues; Childhood Cancer; Psychology, Social
MeSH Terms: conditions — Infertility; Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FERTITOP: 300 patients (15-25 years) from 5 different hospitals (University Hospitals of Nancy, Strasbourg, Reims, Besançon, Dijon (France)) who have finished all cancer treatments for at least 2 years.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will be surveyed through self-administered questionnaires and semidirected interviews with a psychologist
  Other Names: Interview

SUMMARY:
Background: When a cancer is diagnosed in a child, the urgency is to take therapeutic actions. Children and their families face the reality of cancer and the reality of the treatments that, in addition to be overwhelming, might cause infertility. Immediately after the diagnosis, a fertility preservation consultation is proposed to discuss fertility preservation options. In practice, it is often difficult to organize.

Several years after the end of treatments, a second information consultation is proposed to inform about fertility, evaluate the fertility status and propose a second line of Fertility Preservation when possible. The literature reflects a lack of knowledge regarding the degree of fertility-related distress among pediatric cancer patients as well as insufficient tools at the disposal of medical doctors and nurses to discuss about reproduction with children and young adolescents.

Project objective: Understand how young cancer patients and their parents felt about sterility risk at the diagnostic time and now as cured adolescents.

Patients & Methods:

300 patients (15-25 years) from 5 different centers (20 patients per year and per center for 3 years) will be included in this study at the information consultation. They will be surveyed through self-administered questionnaires and semidirected interviews that will 1) retrieve perceptions and emotional being of children during the fertility preservation consultation; 2) assess the decision-making process of parents and family since the fertility preservation consultation through the patient's speech; 3) interview the patients about personal history and experience of cancer and consequences of potential fertility impairment and 4) survey the current experience and projections in the future and evaluate their reaction to the proposition of a second line of Fertility Preservation.

Expected results: what points should the doctor / psychologist discuss with pediatric cancer survivors in response to their fertility stress? and how to do it? for better initial and follow-up care to improve their quality of life after cancer.

ELIGIBILITY:
Inclusion Criteria:

* age between 15 -25
* having been diagnosed with cancer during childhood or adolescence,
* having finished the treatments and being in remission for at least 2 years

Exclusion Criteria:

* Recurrence of cancer at the time of the study
* Lack of cognitive autonomy to be able to agree to participate in the study

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults treated for childhood cancer in one of the five hospital of the Great Est region or France having a follow-up by a pediatric oncologist.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of infertility on psychological health | december 2023
  Patients will report the outcomes of the infertility risks on the questionnaire provided in this study.
  Positive and negative impacts will be questioned.

SECONDARY OUTCOMES:
Develop a decision aid tool for clinicians designed to increase referral for fertility preservation | december 2023
  Using the factors that facilitate or hinder referral to fertility preservation to create a tool for clinicians designed to increase the referral for fertility preservation of children and adolescents with cancer

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - University Hospital of Besançon, Besançon
  - University Hospital of Dijon, Dijon
  - University Hospital of Nancy, France, Nancy
  - University hospital of Reims, Reims
  - University hospital of Strasbourg, Strasbourg